CLINICAL TRIAL: NCT01268670
Title: Adjunctive Oral Analgesia for Laceration Repair: Assessing Pain in a Pediatric Emergency Department
Brief Title: The Addition of Oral Analgesics to LET During Laceration Repair
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is currently suspended due to transition of the investigator.
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Principal Investigator, Heidi Vander Velden, Senior Clinical Research Coordinator, Children's Hospitals and Clinics of Minnesota
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1005-052
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Laceration; Pain
MeSH Terms: conditions — Lacerations; Pain | interventions — Ibuprofen; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Ibuprofen (Active Comparator): Subjects will receive topical LET and oral ibuprofen.
  Interventions: Drug: Ibuprofen
- Oxycodone (Active Comparator): Subjects will receive topical LET and oral oxycodone.
  Interventions: Drug: Oxycodone
- Placebo (Placebo Comparator): Subjects will receive topical LET and oral placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ibuprofen — Subjects will receive topical LET and oral ibuprofen.
  Arms: Ibuprofen
Drug: Oxycodone — Subjects will receive topical LET and oral oxycodone.
  Arms: Oxycodone
Other: Placebo — Subjects will receive topical LET and oral placebo.
  Arms: Placebo

SUMMARY:
Background Approximately 30 million children are treated in emergency departments each year in the United States, of which two to three million are children presenting with lacerations. Topical numbing medication is the standard of care in children with regard to pain control during laceration repair. While topical numbing medications are effective, children often require further pain control during laceration repair in the form of an injected numbing medication, which in itself is painful. No evidence currently exists regarding the concurrent use of oral pain medications to combat laceration procedural pain.

Research Question Does the addition of ibuprofen or oxycodone to lidocaine, epinephrine, and tetracaine (LET) topical anesthetic provide more effective pain control than LET alone during laceration repair?

Design This is a double-blinded, randomized-controlled study.

Methods Subjects in all three groups will receive topical anesthetic. In addition to topical anesthetic, two groups of children will receive either of two oral analgesics, ibuprofen or oxycodone, while the third group will receive a placebo.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking patients
* Patients 4 years of age up to 10 years of age
* Patients seen in the ED needing simple facial laceration repair
* Patients with no chronic medical problems

Exclusion Criteria:

* Any patient who's parent or primary caretaker refuses consent
* Any patient who's parent or primary caretaker needs an interpreter
* Any child with complex laceration(s) or bites
* Any child who has received pain medication at home in response to the facial laceration.
* Children needing procedural sedation
* Children with a known allergy to lidocaine, epinephrine, tetracaine, ibuprofen, or oxycodone
* Patients with known or pre-existing medical conditions where the study protocol cannot be used
* This includes any patient with a medical condition that prevents appropriate use of the pain scale
* It also includes patients with medical conditions that warrant the use of chronic medications

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Pain scores | At Triage, after first suture, and the worst during the procedure
  The use of adjunctive oral analgesics for facial/scalp laceration repair decrease pain scores more effectively than LET alone.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis and Saint Paul, Minnesota, United States